CLINICAL TRIAL: NCT05933200
Title: A Randomized, Double-blind, Multicenter Study to Determine the Effect of Triheptanoin Compared With Even-chain, Medium-chain Triglycerides (MCT) on Major Clinical Events (MCEs) in Pediatric Patients With Long-chain Fatty Acid Oxidation Disorders (LC-FAOD)
Brief Title: A Study to Determine the Effect of Triheptanoin Compared With Even-Chain MCT on MCEs in Pediatric Patients With LC-FAOD
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UX007-CL302; 2022-001539-10 (EudraCT Number); 2023-509809-76-00 (EU CTIS Number)
Record Dates: First submitted 2023-06-27; First posted 2023-07-06 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Long-chain Fatty Acid Oxidation Disorders (LC-FAOD)
Keywords: Carnitine Palmitoyl Transferase (CPT) I Deficiency; Carnitine Palmitoyl Transferase (CPT) II Deficiency; Carnitine/acylcarnitine Translocase (CACT) Deficiency; Very Long Chain Acyl-coenzyme A Dehydrogenase (VLCAD) Deficiency; Long-chain 3-hydroxyacyl-coenzyme A Dehydrogenase (LCHAD) Deficiency; Mitochondrial Trifunctional Protein (TFP) Deficiency
MeSH Terms: conditions — VLCAD deficiency | interventions — triheptanoin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Triheptanoin (Experimental): Participants will be given prescriptions for triheptanoin in mL/day, which will be divided into approximately 4 administrations per day, with precise instructions for administration. Triheptanoin will be titrated up to the first 6 weeks of the study. After titration, the dose is to remain stable for the remainder of the Double-blind Treatment Period. Following the Double-blind Treatment Period, open-label triheptanoin will be provided at participants' current dose during an Open Access Period, if no other options to receive trihepatnoin are available locally.
  Interventions: Drug: Triheptanoin
- MCT (Active Comparator): Participants will be given prescriptions for MCT in mL/day, which will be divided into approximately 4 administrations per day, with precise instructions for administration. MCT will be titrated up to the first 6 weeks of the study. After titration, the dose is to remain stable for the remainder of the Double-blind Treatment Period. Following the Double-blind Treatment Period, open-label triheptanoin will be provided at participants' current dose during an Open Access Period, if no other options to receive trihepatnoin are available locally.
  Interventions: Dietary Supplement: MCT Oil

INTERVENTIONS:
Drug: Triheptanoin — Liquid for oral (PO) or enteral feeding tube administration
  Other Names: UX007; Dojolvi
  Arms: Triheptanoin
Dietary Supplement: MCT Oil — Liquid for oral (PO) or enteral feeding tube administration
  Other Names: Medium-chain Triglyceride
  Arms: MCT

SUMMARY:
The main goal of this study is to evaluate the effects of triheptanoin versus Medium-chain Triglycerides (MCT) on frequency of Major Clinical Events (MCEs).

DETAILED DESCRIPTION:
Participants will be randomly assigned 1:1 to receive triheptanoin or MCT oil. The duration of the study is estimated to be 3.5 to 4 years. The study comprises the following: Screening Period, Baseline (Month 0), Double-blind Treatment Period (including Titration and End of Study Visit), Safety Follow-up Phone Visit, and an Open Access Period.

In addition, a substudy will examine the effect of triheptanoin versus MCT on decreasing liver fat fraction to avoid or improve steatosis in subjects with LC-FAOD. Participants older than 2 years of age at selected sites will be invited to screen for the Liver Substudy.

ELIGIBILITY:
Inclusion Criteria for Main Study:

* Males and females, from 0 (including newborns) to < 18 years of age at time of randomization
* Confirmed diagnosis of LC-FAOD
* Have a caregiver(s) willing and able to assist in all applicable study requirements
* Have a legally authorized representative willing and able to provide written informed consent after the nature of the study has been explained and prior to any research-related procedures, and the study participant to be able to provide age-appropriate written assent
* Have ANY ONE of the following significant clinical manifestations of LC-FAOD:

  * At least 2 in the prior year, or 3 in the prior 2 years, of severe major episodes of metabolic decompensation (eg, hypoglycemia, rhabdomyolysis, or exacerbation of cardiomyopathy, requiring ER/urgent care unit visits or hospitalizations)
  * Recurrent symptomatic hypoglycemia (clinical symptoms of hypoglycemia) requiring intervention
  * Susceptibility to hypoglycemia after short periods of fasting (less than 4 to 12 hours, depending on age)
  * Evidence of functional cardiomyopathy requiring ongoing medical management or clinical manifestation of heart failure
  * Sibling(s) with the same pathogenic variant who presented with MCEs
  * Participant with pathogenic variants that are known or suspected to be associated with absent or severely reduced enzyme activity or with severe disease manifestations.
* From the period following informed consent to 5 days after the last dose of study drug, females of childbearing potential and fertile males must consent to use highly effective contraception. If female, agree not to become pregnant. If male, agree not to father a child or donate sperm

Inclusion Criteria for Liver Substudy:

* Enrollment in the Main Study of Study UX007-CL302
* Age > 2 years
* Liver fat content ≥ 2% and < 20% PDFF as assessed by 1 H-MRS
* Body mass index < 95th percentile
* Able to comply with instructions (remaining still during scan) and requirements (eg, constraints on recent meals, no metallic items or implanted devices in the body, no recent contrast agents) for liver 1 H-MRS scan

Exclusion Criteria for Main Study:

* Enrolled in a clinical study involving concurrent use of an investigational drug product within 30 days before Screening
* Use of a prohibited medication (eg, valproate products or pancreatic lipase inhibitors) within 30 days before Screening, or unwilling to avoid a prohibited medication or other substance that may confound study objectives
* Treatment with triheptanoin within 60 days of Screening
* History of known hypersensitivity to triheptanoin or MCT or its excipients that, in the judgement of the Investigator, places the subject at increased risk for adverse effects
* Caregiver unwilling or unable to sign informed consent, or release of medical records, or follow study procedures
* Have any comorbid conditions, including unstable major organ-system disease(s), that in the opinion of the Investigator places the subject at increased risk of complications, interferes with study participation or compliance, or confounds study objectives or interpretation of results. History of metabolic decompensation(s) with metabolic acidosis, hyperammonemia, and/or liver enzyme elevations does not constitute an exclusion criterion unless in the opinion of the Investigator places the subject at increased risk of complications, interferes with study participation or compliance, or confounds study objectives or interpretation of results.
* Have a diagnosis of pancreatic insufficiency
* Pregnant, breastfeeding, or planning to become pregnant (self or partner) at any time during the study

Exclusion Criteria for Liver Substudy:

* Acute or chronic liver disease other than LC-FAOD that presents with increased risk of liver fat (eg, hepatic cirrhosis, viral toxic or drug hepatitis, diabetes mellitus) and/or metabolic syndrome
* Need for anesthesia/sedation to perform liver 1 H-MRS

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 69 (Actual)
Dates: Start 2023-02-28 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Annualized Event Rate of Major Clinical Events (MCEs) | Up to Year 4

SECONDARY OUTCOMES:
Annualized Duration of MCEs | Up to Year 4
Annualized Hypoglycemic Event-rate Captured as MCEs and At-home Clinical Events (HCEs) | Up to Year 4
Clinical Global Impression of Change [CGI-C] Scale Score | Up to Year 4
Change From Baseline in Left Ventricular Ejection Fraction | Baseline, Up to Year 1
Change From Baseline in Left Ventricular Systolic Volume | Baseline, Up to Year 1
Change From Baseline in Left Ventricular Wall Mass | Baseline, Up to Year 1
Liver Substudy (Single Study Site Only): Change from Baseline to 6 Months in Hepatic Proton Density Fat Fraction (PDFF%), Assessed by 1H-Magnetic Resonance Spectroscopy (1H-MRS) | Baseline, Month 6
Annualized Frequency of Rhabdomyolysis-MCEs and Cardiomyopathy-MCEs | Up to Year 4
Annualized Duration of Rhabdomyolysis-MCEs, Cardiomyopathy-MCEs, and Hypoglycemic-MCEs | Up to Year 4
Change From Baseline in Caregiver-reported Pediatric Quality of Life Inventory (PedsQL) 4.0 Generic Core Scale Score for Participants 2 Years of Age or Older | Up to Year 4
Change From Baseline in PedsQL Infant Scale Score for Participants Ages 1 to <24 Months | Up to Year 4
Survival Time | Up to Year 4
Annualized Hospitalization Days | Up to Year 4
Number of Missed School or Learning Opportunity Days | Up to Year 4
Number of Participants With Treatment-emergent Adverse Events (TEAEs), Serious TEAEs, and Adverse Events of Special Interest (AESIs) | Up to Year 4
Number of Participants With TEAEs and Serious TEAEs Leading to Dose Modifications, Dose Reductions, Treatment Interruptions, Discontinuations From Study Drug, and Discontinuations From the Study | Up to Year 4
Plasma Concentration Levels of Heptanoate | Up to Year 1
Plasma Concentration Levels of Beta Hydroxypentanoate (BHP) | Up to Year 1
Acceptability and Palatability Survey Scores of Triheptanoin Mixed with Oral Liquids | Up to Year 1

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Ultragenyx Pharmaceutical Inc
Locations (15):
- General University Hospital in Prague-GUH (Všeobecná fakultní nemocnice v Praze- VFN), Prague, Czechia
- Universitätsklinikum Freiburg, Freiburg im Breisgau, Germany
- Japan (2):
  - Juntendo University Hospital, Bunkyo City, Tokyo
  - The Jikei University Hospital, Minato, Tokyo
- Poland (2):
  - Instytut Pomnik-Centrum Zdrowia Dziecka, Warsaw, Masovian Voivodeship
  - Gdańksi Uniwersytet Medyczny, Gdansk, Pomeranian Voivodeship
- King Faisal Specialist Hospital & Research Centre, Riyadh, Saudi Arabia
- Spain (3):
  - Sant Joan de Deu Hospital (SJD), Barcelona, Esplugues de Llobregat
  - University Hospital Santiago de Compostela, A Coruña
  - University Hospital 12 de Octubre, Madrid
- Turkey (Türkiye) (5):
  - Cukurova University, Adana
  - Gazi University, Ankara
  - Ege University, Bornova-İzmir
  - Istanbul Universitesi Istanbul Tip Fakultesi Hastanesi, Istanbul
  - Cerrahpasa Medical Faculty, Istanbul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Ultragenyx Patient Advocacy/LC-FAOD Disease Information — https://ultrarareadvocacy.com/conditions-we-study/long-chain-fatty-acid-oxidation-disorders-lc-faod/
- See also: Ultragenyx Transparency Commitment — https://www.ultragenyx.com/our-research/our-clinical-trial-transparency-commitment/